CLINICAL TRIAL: NCT02157909
Title: Daily Wear (DW) Evaluation of Lotrafilcon B in a Modified Design
Brief Title: DW Evaluation of Lotrafilcon B Lenses in a Modified Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C-13-055
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Myopia
Keywords: Lens fit; contact lenses; myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOA Modified (Experimental): Lotrafilcon B sphere modified design contact lenses worn at least 8 hours per day, 5 days per week on a daily wear basis for 7 days.
  Interventions: Device: Lotrafilcon B sphere modified design contact lenses
- AOA (Active Comparator): Lotrafilcon B sphere contact lenses worn at least 8 hours per day, 5 days per week on a daily wear basis for 7 days.
  Interventions: Device: Lotrafilcon B sphere contact lenses

INTERVENTIONS:
Device: Lotrafilcon B sphere modified design contact lenses
  Arms: AOA Modified
Device: Lotrafilcon B sphere contact lenses
  Other Names: AIR OPTIX® AQUA sphere; AOA
  Arms: AOA

SUMMARY:
The purpose of this study is to demonstrate that Lotrafilcon B AIR OPTIX® AQUA sphere modified design lenses are noninferior to Lotrafilcon B AIR OPTIX® AQUA in overall lens fit by comparing the percent of subjects satisfying the "no re-fit" criteria in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent Document;
* Myopic, wear AIR OPTIX® AQUA lenses in the range of -1.00 to -5.00 diopters (D) in both eyes, and willing to comply with the wearing schedule;
* Manifest cylinder less than or equal to 0.75 D;
* Able to achieve best corrected visual acuity (BCVA) of 20/25 (Snellen) or better in each eye at distance;
* Able to achieve distance visual acuity of at least 20/40 in each eye with habitual and study lenses;
* Wearing spherical AIR OPTIX® AQUA lenses in both eyes for at least 3 months (at least 8 hours per day, at least 5 days per week), wearing the habitual lenses for a minimum of 4 hours prior to the baseline study visit, and achieving an acceptable or optimal fit at baseline visit with habitual lenses in both eyes;
* Other protocol-defined criteria may apply.

Exclusion Criteria:

* Current soft contact lens wearer who regularly sleeps in lenses (1 or more nights per week);
* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear within 6 months prior to enrollment;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated including any use of topical ocular medications that would require instillation during contact lens wear;
* History of herpetic keratitis;
* History of corneal or refractive surgery or irregular cornea;
* A pathologically dry eye that precludes contact lens wear;
* Monocular (only one eye with functional vision);
* Monovision correction;
* History of intolerance or hypersensitivity to any component of the test articles or associated materials;
* Concurrent participation in a contact lens or contact lens care product clinical trial or within the previous 30 days;
* Eye injury or ocular or intra-ocular surgery within 6 months prior to enrollment;
* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the study lenses or affect the results of this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, Vision Care, GCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 study centers located in the US.
Pre-assignment Details: Of the 134 enrolled, 2 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (132).
Groups:
- AOA Modified: Modified design contact lenses worn at least 8 hours per day, 5 days per week on a daily wear basis for 7 days
- AOA Sphere: Sphere contact lenses worn at least 8 hours per day, 5 days per week on a daily wear basis for 7 days
Period: Overall Study
Arm/Group | AOA Modified | AOA Sphere
Started | 66 | 66
Completed | 66 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | AOA Modified | AOA Sphere | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (9.5) | 31.3 (9.8) | 30.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 95
  Male | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Satisfying the 'no Re-fit' Criteria in Both Eyes
Description: With the contact lens on eye, the investigator assessed the lens fit immediately post-blink and following lower lid margin push-up with the lower lid using a 5-point scale, where -2 = Unacceptably tight (reduced movement, unacceptable), -1 = Acceptably tight (reduced movement, acceptable), 0 = Optimal fit / movement, +1 = Acceptably loose (excessive movement, acceptable), and +2 = Unacceptably loose (excessive movement, unacceptable). To meet the definition of "no re-fit," an eye had to have an acceptable or optimal overall lens fit with the study lens, as well as be within 1 grade of the overall lens fit assessed with the habitual lens at baseline. Proportion of subjects is reported as a percentage.
Time Frame: Dispense (Day 0), Week 1
Population: This analysis population includes all randomized and treated subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | AOA Modified | AOA Sphere
Number analyzed (Participants) | 66 | 66
percentage of subjects
  Dispense (Day 0) | 100.0 | 100.0
  Week 1 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (June 2014 - July 2014). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device (test article) and control article.
Groups:
- Pre-treatment: Includes all subjects / eyes prior to the exposure to the investigational or control products
- AOA Modified: Includes all subjects / eyes exposed to AOA Modified lenses
- AOA Sphere: Includes all subjects / eyes exposed to AOA Sphere lenses
Arm/Group | Pre-treatment | AOA Modified | AOA Sphere
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/134 | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.